CLINICAL TRIAL: NCT07047508
Title: A Non-interventional Study of the Effectiveness and Safety Outcomes in Patients With Heart Failure and Preserved Ejection Fraction (HFpEF) Initiating Jardiance in China: A Sub-study of the Post-marketing Study of Jardiance Among Patients With Heart Failure in China
Brief Title: Real-world Study to Describe the Effectiveness and Safety Outcomes of Jardiance in Chinese Patients With Heart Failure and Preserved Ejection Fraction
Status: Not yet recruiting | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0313
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure; Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart failure and preserved ejection fraction patients

SUMMARY:
The main objective of the study is to describe the effectiveness and safety outcomes among Chinese hospitalized heart failure with preserved ejection fraction (HFpEF) patients initiating Jardiance® in the real-world setting.

ELIGIBILITY:
Inclusion criteria:

* At least 18 years of age
* At least 6 months of data prior to the index date
* Left ventricular ejection fraction (LVEF) > 40 %
* N-terminal Pro-B-type natriuretic peptide (NT-proBNP) > 125 pg/mL or brain natriuretic peptide (BNP) ≥ 35 pg/mL
* At least 1 diagnosis of Heart failure with preserved ejection fraction (HFpEF) or Heart failure with mid-range ejection fraction (HFmrEF) or chronic heart failure (CHF) at baseline during the look-back period (on or prior to the index date)
* New users of Jardiance® (initiating Jardiance® on or after March 1st, 2023, and without any record of Jardiance® prescription during the look-back period)
* Body Mass Index (BMI) <45 kg/m2

Exclusion criteria:

-Patients treated with any other sodium-glucose cotransporter-2 inhibitors (SGLT2i) on the index date or during the look-back period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chines patients with a heart failure and preserved ejection fraction (HFpEF) diagnosis who initiate Jardiance® after 1st of March 2023
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of the composite outcome of HHF (the first HHF after the index date) or CV death | up to 2.5 years
  HHF=Hospitalization for Heart Failure CV=cardiovascular

SECONDARY OUTCOMES:
Incidence of CV death | up to 2.5 years
Incidence of the HHF (the first HHF after the index date) | up to 2.5 years
Occurrence of death from any cause | up to 2.5 years

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com